CLINICAL TRIAL: NCT06809127
Title: Etude de la plasticité cérébrale et de la Reconnaissance Des émotions en magnétoencéphalographie Chez Les Patients paralysés Faciaux Avant et après réhabilitation Motrice de la Face
Brief Title: Brain Plasticity and Emotion Recognition in Patients With Facial Palsy Before & After Surgical Rehabilitation: MEG Study
Acronym: FACE_REHAB_MEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Fondation des Gueules Cassées (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C16-70; 2016-A01861-50 (Registry Identifier: IDRCB)
Record Dates: First submitted 2017-05-03; First posted 2025-02-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Facial Palsy; Surgery
Keywords: facial palsy; brain plasticity; motor cortex; emotion; MEG
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral tasks with MEG recording (Other): 1. MOTOR TASK: Five types of simple movements will be performed: eye blinks, smiling, tongue protraction, teeth greeting, index flexion. A total of 120 movements of each type will be performed in a set of five blocks interspersed with short breaks.
  2. EMOTION RECOGNITION TASK: Four emotional expressions will be presented: happiness, anger, sadness, and neutral expression. A total of 320 face stimuli will be presented in 5 blocks interspersed with short breaks. Occasional target faces displaying a suprised expression will be added. The patient's task will be to report the occurrence of those faces by pressing a button in his/her dominant hand.
  Interventions: Device: Behavioral tasks with MEG recording

INTERVENTIONS:
Device: Behavioral tasks with MEG recording — The patients will undergo two visits, during which MEG will be recorded in two types of behavioral tasks: motor task and emotion recognition task. One visit will take place before surgery. The second visit will take place after the surgical intervention and the face motor rehabilitation, 3 to 18 months after the 1st visit.

SUMMARY:
Facial palsy (of one hemiface) affects the sensorimotor representation of the face of the patients, and possibly also their mental representation of emotional facial expressions. Three surgical techniques are performed to rehabilitate the face motricity in patients with severe facial palsy: Facio-facial anastomosis (AFF), Hypoglosso-facial anastomosis (AHF), and Lengthening temporalis myoplasty (LTM). Our objective is to study brain plasticity and facial emotion recognition in patients with facial palsy before and after surgical rehabilitation, using non invasive magnetoencephalography (MEG) recording during motor and emotion recognition tasks.

DETAILED DESCRIPTION:
Facial palsy (of one hemiface) affects the sensorimotor representation of the face of the patients, and possibly also their mental representation of emotional facial expressions. Patients with severe facial palsy can benefit from surgical rehabilitation, allowing them to recover the motor and expressive function of the face. Three surgical techniques are performed to rehabilitate facial palsy: Facio-facial anastomosis (AFF), Hypoglosso-facial anastomosis (AHF), and Lengthening temporalis myoplasty (LTM). Prinicipal objective is to study brain plasticity and facial emotion recognition in patients with facial palsy before and after surgical rehabilitation. For this, the investigators will use magnetoencephalography (MEG), which is a non-invasive brain imaging method with high temporal and good spatial resolution.

1. First objective is to characterize the brain plasticity at a global level, independently of the surgical technique used. The investigators will use simple motor tasks consisting in performing different facial movements and a control index flexion task to examine the cortical plasticity associated with the restauration of the motor and expressive function of the face in patients with facial palsy.
2. Second objective is to examine if the brain magnetic responses associated with the recognition of emotional faces are modified in the paralyzed patients. The investigators will study the brain responses to angry, sad, happy, and neutral faces in a simple emotion recognition task.

Twenty patients with facial palsy will be included in the study. They will undergo two visits, during which MEG will be recorded in two types of tasks: motor task and emotion recognition task (see below). One visit will take place before surgery. The second visit will take place after the surgical intervention and the face motor rehabilitation, 3 to 18 months after the 1st visit.

MOTOR TASK: The motor task will comprise 5 types of simple movements: eye blinks, smiling, tongue protraction, teeth greeting, index flexion. These movements will be performed repetitively - at a pace of about 1 movement every 2 second - in separate, randomly alternating, blocks of 24 movements of each type, for a total of 120 movements of each type.

EMOTION RECOGNITION TASK: A total of 320 faces will be presented to the patients. The faces will be distributed in 5 blocks of 16 different faces (8 male, 8 female), displaying each of 4 emotional expressions: happiness, anger, sadness, and neutral expression. Occasional suprised target faces will be added. The patient's task will be to report the occurrence of those faces by pressing a button in his/her dominant hand. The stimuli will be presented in random order in each block.

The investogators will analyze neuromagnetic activities at the sensor and source levels during the motor tasks (primary objective) and in response to the faces (secondary objective).

ELIGIBILITY:
Inclusion Criteria:

* No history of psychiatric illness
* Severe facial palsy (V or VI grade on House and Brackman scale)
* No evolutive neurologic pathology beside the lesion of the VIIth nerve
* Signature of informed consent
* Being a member of, or beneficiary of, a social security scheme

Exclusion Criteria:

* Evolutive neurological disease outside the lesion of the VIIth nerve
* General pathology leading to neuropathy
* Person unable to express his/her consent
* Adult under a legal protection measure
* Adult deprived of liberty by judicial or administrative decision.
* Adult participating in another research protocol involving the human person or subjected to a period of exclusion from another research
* Claustrophobia
* Implants or metallic objects (including eyeglasses) that are susceptible to pertrubate the MEG signal
* Treatment with known action on the central nervous system (Excessive recreational use of psychotropic drugs, ongoing benzodiazepine therapy)
* For the patients who will undergo a complementary structural MRI for MEG source localisation, additional exclusion criteria are the contraindications to MRI (including: pacemaker or neurosensitive stimulator or implanted defibrillator, anevrism or vascular malformation of the brain, cochlear implants, ferromagnetic objects or prosthesis in the eyes or brain, mechanical heart valve prosthesis, permanent eye makeup; pregnant or nursing women)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Magnetoencephalography (MEG) activities during facial motor tasks | between 3 and 18 months
  Magnetoencephalography (MEG) activities during the motor tasks

SECONDARY OUTCOMES:
Magnetoencephalography (MEG) activities in reponse to emotional faces | between 3 and 18 months
  Magnetoencephalography (MEG) activities in reponse to sad, angry, happy, and neutral faces during the facial emotion recognition task

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric TANKERE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Frederic TANKERE, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foirest C, Gatignol P, Bernat I, Lamas G, Tankere F. [Lengthening temporalis myoplasty for facial palsy reanimation after parotid surgery]. Rev Laryngol Otol Rhinol (Bord). 2013;134(4-5):259-65. French. PMID 25252584
- [Background] Garmi R, Labbe D, Coskun O, Compere JF, Benateau H. Lengthening temporalis myoplasty and brain plasticity: a functional magnetic resonance imaging study. Ann Chir Plast Esthet. 2013 Aug;58(4):271-6. doi: 10.1016/j.anplas.2013.03.002. Epub 2013 Apr 23. PMID 23623628
- [Background] Leonetti JP, Anderson DE, Marzo SJ, Origitano TC, Petruzzelli GJ. Intratemporal Grafting of the Facial Nerve following Lateral Skull Base Tumor Resection. Skull Base. 2007 May;17(3):181-6. doi: 10.1055/s-2007-977464. PMID 17973031
- [Background] Memarian N, Ferrari P, Macdonald MJ, Cheyne D, De Nil LF, Pang EW. Cortical activity during speech and non-speech oromotor tasks: a magnetoencephalography (MEG) study. Neurosci Lett. 2012 Oct 3;527(1):34-9. doi: 10.1016/j.neulet.2012.08.030. Epub 2012 Aug 25. PMID 22926020
- [Background] Miki K, Kakigi R. Magnetoencephalographic study on facial movements. Front Hum Neurosci. 2014 Jul 29;8:550. doi: 10.3389/fnhum.2014.00550. eCollection 2014. PMID 25120453
- [Background] Nakahara H, Nakasato N, Kanno A, Murayama S, Hatanaka K, Itoh H, Yoshimoto T. Somatosensory-evoked fields for gingiva, lip, and tongue. J Dent Res. 2004 Apr;83(4):307-11. doi: 10.1177/154405910408300407. PMID 15044504
- [Background] Nakamura A, Yamada T, Goto A, Kato T, Ito K, Abe Y, Kachi T, Kakigi R. Somatosensory homunculus as drawn by MEG. Neuroimage. 1998 May;7(4 Pt 1):377-86. doi: 10.1006/nimg.1998.0332. PMID 9626677
- [Background] Nakasato N, Itoh H, Hatanaka K, Nakahara H, Kanno A, Yoshimoto T. Movement-related magnetic fields to tongue protrusion. Neuroimage. 2001 Oct;14(4):924-35. doi: 10.1006/nimg.2001.0881. PMID 11554811
- [Background] Rijntjes M, Tegenthoff M, Liepert J, Leonhardt G, Kotterba S, Muller S, Kiebel S, Malin JP, Diener HC, Weiller C. Cortical reorganization in patients with facial palsy. Ann Neurol. 1997 May;41(5):621-30. doi: 10.1002/ana.410410511. PMID 9153524
- [Background] Salmelin R, Sams M. Motor cortex involvement during verbal versus non-verbal lip and tongue movements. Hum Brain Mapp. 2002 Jun;16(2):81-91. doi: 10.1002/hbm.10031. PMID 11954058
- [Background] Suzuki M, Wasaka T, Inui K, Kakigi R. Reappraisal of field dynamics of motor cortex during self-paced finger movements. Brain Behav. 2013 Nov;3(6):747-62. doi: 10.1002/brb3.186. Epub 2013 Oct 17. PMID 24363977
- [Background] Tankere F, Bernat I, Vitte E, Lamas G, Soudant J, Maisonobe T, Bouche P, Fournier E, Willer JC. [The hypolossal-facial anastomosis in man. A model for studying peripheral and central nervous system plasticity]. Rev Med Liege. 2004;59 Suppl 1:91-103. French. PMID 15244163
- [Background] Vvedensky VL, Prokofyev AO. Timing of Cortical Events Preceding Voluntary Movement. Neural Comput. 2016 Feb;28(2):286-304. doi: 10.1162/NECO_a_00802. Epub 2015 Dec 14. PMID 26654207
- [Background] Willer JC, Tankere F, Maisonobe T, Bernat I, Lamas G, Soudant J, Vitte E, Bouche P, Fournier E. Hypoglossal-facial anastomosis induced central plastic changes in the blink reflex circuitry. Mov Disord. 2002;17 Suppl 2:S53-7. doi: 10.1002/mds.10060. No abstract available. PMID 11836756
- [Background] Yang TT, Gallen CC, Schwartz BJ, Bloom FE. Noninvasive somatosensory homunculus mapping in humans by using a large-array biomagnetometer. Proc Natl Acad Sci U S A. 1993 Apr 1;90(7):3098-102. doi: 10.1073/pnas.90.7.3098. PMID 8464929
- [Result] Hervochon R, Chaumon M, Ziri D, Foirest C, Schwartz D, George N, Tankere F. Cerebral Plasticity after Lengthening Temporalis Myoplasty in Facial Palsy: A Magnetoencephalography Study. Facial Plast Surg Aesthet Med. 2025 Mar-Apr;27(2):145-147. doi: 10.1089/fpsam.2023.0235. Epub 2024 May 13. No abstract available. PMID 38738297